CLINICAL TRIAL: NCT07040644
Title: A Multi-center, Open-label, Randomized, Phase II Trial of Sacituzumab Govitecan Plus Toripalimab Versus Toripalimab Plus Nab-Paclitaxel as First-line Therapy in Patients With Unresectable, Locally Advanced or Metastatic Triple-Negative Breast Cancer
Brief Title: A Study of Sacituzumab Govitecan Plus Toripalimab Versus Toripalimab Plus Nab-Paclitaxel in PD-L1 Positive Advanced TNBC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO-US-979-7331
Record Dates: First submitted 2025-06-19; First posted 2025-06-27 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-05

CONDITIONS: Triple Negative Breast Neoplasms
Keywords: PD-L1 Positive; Sacituzumab Govitecan; Toripalimab; Nab-Paclitaxel; Advanced Breast Cancer; Metastatic TNBC; Randomized Controlled Trial; Progression-Free Survival
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — sacituzumab govitecan; toripalimab; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SG plus Toripalimab (Experimental): Participants will receive sacituzumab govitecan at 10 mg/kg via IV infusion on Days 1 and 8 of each 21-day cycle, and toripalimab at 240 mg via IV infusion on Day 1 of each 21-day cycle. Treatment continues until disease progression, unacceptable toxicity, or withdrawal.
  Interventions: Drug: Sacituzumab Govitecan (SG); Drug: Toripalimab
- Nab-Paclitaxel plus Toripalimab (Active Comparator): Participants will receive toripalimab at 240 mg via IV infusion on Day 1 of each 21-day cycle, and nab-paclitaxel at 125 mg/m² via IV infusion on Days 1 and 8 of each cycle. Treatment continues until disease progression, unacceptable toxicity, or withdrawal.
  Interventions: Drug: Toripalimab; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Sacituzumab Govitecan (SG) — Sacituzumab govitecan will be administered at 10 mg/kg via intravenous infusion on Days 1 and 8 of each 21-day cycle. The treatment continues until disease progression, unacceptable toxicity, or patient withdrawal.
  Arms: SG plus Toripalimab
Drug: Toripalimab — Toripalimab will be administered at a fixed dose of 240 mg via intravenous infusion on Day 1 of each 21-day cycle. Treatment continues until disease progression, unacceptable toxicity, or patient withdrawal.
Drug: Nab-paclitaxel — Nab-paclitaxel will be administered at 125 mg/m² via intravenous infusion on Days 1 and 8 of each 21-day cycle. Treatment continues until disease progression, unacceptable toxicity, or patient withdrawal.
  Arms: Nab-Paclitaxel plus Toripalimab

SUMMARY:
This is a multicenter, open-label, randomized phase II trial evaluating the efficacy and safety of sacituzumab govitecan plus toripalimab versus toripalimab plus nab-paclitaxel in patients with previously untreated, unresectable, locally advanced or metastatic triple-negative breast cancer (TNBC) that is PD-L1 positive.

Eligible patients will be randomized in a 1:1 ratio to receive either sacituzumab govitecan plus toripalimab or toripalimab plus nab-paclitaxel. Tumor response will be assessed by investigators according to RECIST v1.1 at baseline, every 6 weeks during the first year, and every 12 weeks thereafter.

The primary objective is to evaluate progression-free survival (PFS). Secondary endpoints include overall survival (OS), objective response rate (ORR), duration of response (DOR), time to response (TTR), and safety profile according to NCI-CTCAE v5.0.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥18 years.
* Histologically or cytologically confirmed triple-negative breast cancer (TNBC).
* Unresectable locally advanced or metastatic disease.
* PD-L1 positive (CPS ≥1 as assessed by central laboratory).
* No prior systemic treatment for advanced or metastatic TNBC.
* Measurable disease per RECIST v1.1.
* ECOG performance status of 0 or 1.
* Adequate hematologic, hepatic, and renal function.
* Willingness to provide informed consent.

Exclusion Criteria:

* Prior treatment with any anti-PD-1, anti-PD-L1, or anti-CTLA-4 antibodies.
* Known active central nervous system metastases.
* Active autoimmune disease or history of autoimmune disorders requiring systemic treatment.
* Active infection requiring systemic therapy.
* Pregnancy or lactation.
* Other active malignancies requiring treatment within the past 5 years.
* History of severe hypersensitivity reactions to study drugs.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From randomization until disease progression or death, assessed up to 36 months
  Progression-Free Survival (PFS) is defined as the time from randomization to the first occurrence of disease progression or death from any cause, whichever occurs first, as assessed by investigators based on RECIST version 1.1 criteria.

SECONDARY OUTCOMES:
Overall Survival (OS) | From randomization until death, assessed up to 48 months
  Overall Survival (OS) is defined as the time from randomization to death from any cause. The event will be recorded regardless of cause and assessed continuously until the end of study follow-up.
Objective Response Rate (ORR) | From first dose to first confirmed response, assessed up to 36 months
  Objective Response Rate (ORR) is defined as the proportion of patients who achieve a complete response (CR) or partial response (PR), confirmed at least 4 weeks after the initial response, as assessed by investigators according to RECIST version 1.1 criteria.
Duration of Response (DOR) | From first response until progression or death, assessed up to 36 months
  Duration of Response (DOR) is defined as the time from the first documentation of complete response (CR) or partial response (PR) until disease progression or death from any cause, whichever occurs first, as assessed by investigators according to RECIST version 1.1 criteria.
Time to Response (TTR) | From randomization to first response, assessed up to 36 months
  Time to Response (TTR) is defined as the time from randomization to the first documentation of complete response (CR) or partial response (PR), as assessed by investigators according to RECIST version 1.1 criteria.
Incidence of Adverse Events and Serious Adverse Events | From first dose until 30 days after last dose
  Incidence, type, and severity of adverse events (AEs) and serious adverse events (SAEs) will be assessed from the first dose through 30 days after the last dose, and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China